CLINICAL TRIAL: NCT03115450
Title: Comparative Analysis of Pupilometer and Ultrasound Assessment of Optic Nerve Sheath Diameter in Estimating Intracranial Pressure (ICP)
Brief Title: Comparison of Pupilometer and Ultrasound of Optic Nerve Sheath Diameter in Estimating Intracranial Pressure (ICP)
Acronym: CUSPICP
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Ronak Raval, Assistant Professor, Loma Linda University
Other Study IDs: 5170065
Record Dates: First submitted 2017-03-27; First posted 2017-04-14 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Intracranial Hemorrhages; Brain Injuries; Subarachnoid Hemorrhage; Ischemic Stroke; Stroke
Keywords: External ventricular drain (EVD); Placement of Bolt
MeSH Terms: conditions — Intracranial Hemorrhages; Brain Injuries; Subarachnoid Hemorrhage; Ischemic Stroke; Stroke | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Ultrasound — Type of imaging technology to look at organs and structures inside the body
Device: Pupilometer — A device that measures pupil size and how it changes.

SUMMARY:
The purpose of this investigator-initiated study is to compare the use of pupilometer and ultrasound assessment of optic nerve sheath diameter in predicting the ICP and to see if there is a value that could be used to indicate elevated ICP with either modality as these numbers are inconsistent throughout the literature. Patients that have either an external ventricular drain (EVD) or bolt placed will be enrolled in the study. After the EVD and bolt are placed the patient will undergo pupilometer examination (standard of care) followed by ultrasound assessment of the optic nerve sheath diameter (ONSD). The three values will be recorded. The same patient may have multiple readings performed if there is a change in ICP either spontaneously or due to intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Intracranial pathology requiring either EVD or bolt placement for ICP measurement

Exclusion Criteria:

* Known disorder of lens or orbit including but not limited to glaucoma, cataract, blindness, lens implants.
* Patients unable to close eyelids as this would increase risk of corneal abrasion from ultrasound probe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults that have intracranial pathology requiring either EVD or bolt placement for measuring ICP.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Measurement of Optic Nerve Sheath Diameter (ONSD) and corresponding intracranial pressure (ICP). | 1 day of ONSD examination
  Analysis of varying ONSD and pupillometer readings to concurrent ICP

SECONDARY OUTCOMES:
Measurement of Pupillometer reading and corresponding intracranial pressure (ICP). | 1 day per nursing protocol (standard of care)
  Comparison of Neurological Pupil index (NPi) in both eye and concurrent ICP

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

REFERENCES:
- [Background] Chen JW, Gombart ZJ, Rogers S, Gardiner SK, Cecil S, Bullock RM. Pupillary reactivity as an early indicator of increased intracranial pressure: The introduction of the Neurological Pupil index. Surg Neurol Int. 2011;2:82. doi: 10.4103/2152-7806.82248. Epub 2011 Jun 21. PMID 21748035
- [Background] Park JG, Moon CT, Park DS, Song SW. Clinical Utility of an Automated Pupillometer in Patients with Acute Brain Lesion. J Korean Neurosurg Soc. 2015 Oct;58(4):363-7. doi: 10.3340/jkns.2015.58.4.363. Epub 2015 Oct 30. PMID 26587191
- [Background] Taylor WR, Chen JW, Meltzer H, Gennarelli TA, Kelbch C, Knowlton S, Richardson J, Lutch MJ, Farin A, Hults KN, Marshall LF. Quantitative pupillometry, a new technology: normative data and preliminary observations in patients with acute head injury. Technical note. J Neurosurg. 2003 Jan;98(1):205-13. doi: 10.3171/jns.2003.98.1.0205. PMID 12546375
- [Background] Fountas KN, Kapsalaki EZ, Machinis TG, Boev AN, Robinson JS, Troup EC. Clinical implications of quantitative infrared pupillometry in neurosurgical patients. Neurocrit Care. 2006;5(1):55-60. doi: 10.1385/NCC:5:1:55. PMID 16960298
- [Background] Meeker M, Du R, Bacchetti P, Privitera CM, Larson MD, Holland MC, Manley G. Pupil examination: validity and clinical utility of an automated pupillometer. J Neurosci Nurs. 2005 Feb;37(1):34-40. PMID 15794443
- [Background] Shirodkar CG, Munta K, Rao SM, Mahesh MU. Correlation of measurement of optic nerve sheath diameter using ultrasound with magnetic resonance imaging. Indian J Crit Care Med. 2015 Aug;19(8):466-70. doi: 10.4103/0972-5229.162465. PMID 26321806
- [Background] Wroblewski JT, Fadda E, Mazzetta J, Lazarewicz JW, Costa E. Glycine and D-serine act as positive modulators of signal transduction at N-methyl-D-aspartate sensitive glutamate receptors in cultured cerebellar granule cells. Neuropharmacology. 1989 May;28(5):447-52. doi: 10.1016/0028-3908(89)90077-4. PMID 2542835
- [Background] Kimberly HH, Shah S, Marill K, Noble V. Correlation of optic nerve sheath diameter with direct measurement of intracranial pressure. Acad Emerg Med. 2008 Feb;15(2):201-4. doi: 10.1111/j.1553-2712.2007.00031.x. PMID 18275454